CLINICAL TRIAL: NCT00484250
Title: Study of Metronidazole and Doxycycline to Treat Oral Lichen Planus and to Compare Their Efficacy With Each Other
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mashhad University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 240
Record Dates: First submitted 2007-06-07; First posted 2007-06-08 (Estimated); Last update posted 2007-06-11 (Estimated); Status verified 2007-06

CONDITIONS: Oral Lichen Planus
Keywords: Oral Lichen Planus; Metronidazole; Doxycycline
MeSH Terms: conditions — Lichen Planus, Oral | interventions — Metronidazole; Doxycycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: metronidazole,doxycycline

SUMMARY:
Oral lichen planus (OLP) is a chronic inflammatory disorder which causes local irritation,discomfort and subsequent poor dentition and discomfort in eating . Various treatments have been suggested for OLP but their results are unsatisfactory .Despite the fact that steroids have been the main therapeutic choice for many years,some researches have been done regarding the efficacy of other medication such as metronidazole and doxycycline.The purpose of this study is to determine whether metronidazole and doxycycline are effective in the treatment of oral lichen planus and to compare their efficacy with each other.

ELIGIBILITY:
Inclusion Criteria:

* a biopsy-proven untreated OLP of every type with no symptom.

Exclusion Criteria:

* pregnancy, presence of dysplasia in lesions,unilateral lesion suspected lichenoid reaction,history of drinking alcohol in at least 1 month prior to the study, smoking, systemic disease, use of systemic medications and hypersensitivity to the metronidazole and doxycycline.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-09; Study Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arash Mansourian, DDS,MS, Study Chair — Tehran University of Medical Sciences; Majid Sanatkhani, DDS,MS, Study Director — Mashhad University of Medical Sciences; Fatemeh Momen Heravi, Principal Investigator — Tehran University of Medical Sciences
Locations (1):
- Mashhad University Of Medical Sciences(Dentistry School), Mashhad, Khorasan, Iran

REFERENCES:
- See also: Related Info — http://www.emedicine.com/derm/topic663.htm